CLINICAL TRIAL: NCT01962506
Title: Diagnostic Utility of Copeptin in Addition to High-sensitivity Cardiac Troponin for the Early Diagnosis of Non-ST-Elevation Acute Coronary Syndromes - The COPACS Study
Brief Title: Diagnostic Utility of Copeptin in Addition to High-sensitivity Cardiac Troponin for the Early Diagnosis of NSTE-ACS
Acronym: COPACS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: G. d'Annunzio University (Other)
Responsible Party: Principal Investigator, Fabrizio Ricci, MD, Fabrizio Ricci, MD, G. d'Annunzio University
Other Study IDs: COPACS13
Record Dates: First submitted 2013-10-10; First posted 2013-10-14 (Estimated); Last update posted 2013-10-14 (Estimated); Status verified 2013-10

CONDITIONS: Chest Pain
Keywords: Chest pain; Copeptin; High-sensitivity cardiac troponin; Non-ST-Elevation (NSTE) - ACS
MeSH Terms: conditions — Chest Pain; Diabetes Insipidus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Rapid and reliable exclusion of acute myocardial infarction (AMI) during an emergency department (ED) triage is a major unmet clinical need. We aimed at verifying the non-inferiority of a single-sampling strategy of hs-cTn and copeptin compared with the dual hs-cTn sampling for the early diagnosis of Non-ST-Elevation Acute Coronary Syndromes (NSTE-ACS) versus Non Coronary Chest Pain (NCCP) in a selected cohort of consecutive patients admitted at the Emergency Department.

DETAILED DESCRIPTION:
The evaluation of chest pain patients in the emergency department remains a costly and difficult challenge, because a large proportion of them do not suffer from an acute coronary syndrome (ACS). The adequate ruling out of ACS in patients with chest pain is crucial, as the erroneous discharge of a patient with ACS is associated with a high risk of cardiac events. Rapid assessment of these patients is critical to direct further diagnostic and therapeutic strategies. Electrocardiography (ECG) and cardiac troponin (cTn) are the current diagnostic cornerstones and complement clinical assessment in current AMI guidelines1. They allow to rule in an acute myocardial infarction (AMI) within the first 3 hours after presentation in the majority of patients and offer the opportunity to initiate appropriate, evidence-based treatment. The vast majority of patients presenting to the Emergency Department (ED) with suspected AMI, however, finally prove not to have AMI. The current process of ruling out AMI is time-consuming and expensive. One fourth to one-third of patients with AMI present without significant ECG changes indicative of acute ischemia; therefore, the ECG is of little help to rule out AMI, especially in the setting of non-ST elevation ACS (NSTE-ACS). High-sensitivity (hs)-cTn assays have been developed recently, enabling measurements of concentrations that are ∼10-fold lower than those previously measurable. Recent studies have confirmed the increased accuracy of these high-sensitivity assays compared with conventional assays in the early detection of AMI and in the safely ruling in or out of coronary causes of chest pain. However, concerns have been raised about a possible specificity deficit with these new assays. In addition, a second measurement of hs-cTn may be warranted in order to increase the accuracy of the assay.

Copeptin, the C-terminal part of the vasopressin pro-hormone, and a marker of acute endogenous stress, has been demonstrated to be useful for a more rapid ruling out of acute myocardial infarction. Current evidence for the diagnostic validity and performance of a combination of high sensitivity-cardiac troponin and copeptin is limited and controversial. A Bayesian probabilistic approach is likely to be the correct way to evaluate the possible incremental value of copeptin in the detection of ACS. Thus, we aim at prospectively evaluating the diagnostic accuracy of copeptin, hs-cTn, CK-MB and myoglobin, alone or in combination with hs-cTn, for the early diagnosis and ruling out of Non-ST-Elevation (NSTE) ACS versus non-cardiac causes of chest pain in a selected cohort of Emergency Department (ED) chest pain patients according to their pre-test probability, as assessed through a combination of two validated clinical risk score systems (i.e. Chest Pain Score and TIMI Risk Score).

ELIGIBILITY:
Inclusion Criteria:

* Chest pain duration > 5 minutes at rest or upon minimal exertion
* Chest pain onset < 6 hours
* Non-traumatic chest pain

Exclusion Criteria:

* Cardiac arrest
* STEMI
* New left bundle branch block

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the Emergency Department.
Sampling Method: Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2012-12; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Non-inferiority of a single-sampling strategy of hs-cTn and copeptin compared with the dual hs-cTn sampling for the early diagnosis of NSTE-ACS in a selected cohort of consecutive patients admitted at the Emergency Department. | On admission to the Emergency Department
  We aimed at verifying the hypothesis that diagnostic efficiency of the combination of copeptin and hs-cTn on admission would be non-inferior with respect to the 3 hours interval hs-cTn serial sampling for the early diagnosis or ruling out of NSTE-ACS versus non cardiac chest pain in a selected cohort of consecutive ED chest pain patients. According to current international guidelines we selected a 20% difference between serial hscTn levels to establish the diagnosis of myocardial infarction, since the change represented twice the recommended maximum imprecision (a coefficient of variation of 10%).

CONTACTS AND LOCATIONS:
Overall Officials: Fabrizio Ricci, Principal Investigator — Institute of Cardiology and Center of Excellence on Aging, "G. D'Annunzio" University, Chieti, Italy
Locations (1):
- Ospedale Clinicizzato SS. Annunziata, Chieti, Chieti, Italy

REFERENCES:
- [Derived] Ricci F, Di Scala R, Massacesi C, Di Nicola M, Cremonese G, De Pace D, Rossi S, Griffo I, Cataldo I, Martinotti S, Rotondo D, Jaffe AS, Zimarino M, De Caterina R. Ultra-Sensitive Copeptin and Cardiac Troponin in Diagnosing Non-ST-Segment Elevation Acute Coronary Syndromes--The COPACS Study. Am J Med. 2016 Jan;129(1):105-14. doi: 10.1016/j.amjmed.2015.06.033. Epub 2015 Jul 11. PMID 26169889